CLINICAL TRIAL: NCT06740357
Title: Implementation of a Tumor Response Assessment Program Integrating Shared Medical Decision Making Into the Organ Preservation Strategy for Rectal Cancer Patients: Phase III Randomized - Multicenter
Brief Title: Implementation of a Tumor Response Assessment Program Integrating the Shared Medical Decision Into the Organ Preservation Strategy for Rectal Cancer Patients
Acronym: EVAREC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DROUILLARD PHRCK 2023-2
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Tumor response monitoring program with shared decision-making (Experimental)
  Interventions: Other: Tumor response monitoring program; Other: Shared decision-making; Other: Follow-up
- Control: Standard assessment of tumor response (validated in the GRECCAR 2 trial - Lancet 2017) (Active Comparator)
  Interventions: Other: Standard evaluation of tumor response; Other: Decision-making according to national recommendations; Other: Follow-up

INTERVENTIONS:
Other: Tumor response monitoring program — three steps of tumor response evaluation (STEP 1 at 2 months, STEP 2 at 4 months, STEP 3 at 6 months after completion of neoadjuvant treatment): STEP 1: digital rectal examination, pelvic MRI, rectoscopy, TAP scan STEP 2: DRE, pelvic MRI, rectoscopy STEP 3: DRE, pelvic MRI, rectoscopy, TAP or PET scan
  Arms: Experimental: Tumor response monitoring program with shared decision-making
Other: Standard evaluation of tumor response — Assessment at 2 months (+/- 7 days) after neoadjuvant treatment: digital rectal exam, pelvic MRI, rectoscopy, TAP scan
  Arms: Control: Standard assessment of tumor response (validated in the GRECCAR 2 trial - Lancet 2017)
Other: Shared decision-making — At each stage of the monitoring program and depending on the clinical and oncological results, the decision to preserve the rectum will be discussed with the patient according to a shared-decision program.
  Arms: Experimental: Tumor response monitoring program with shared decision-making
Other: Decision-making according to national recommendations — The decision to preserve the rectum is based on assessment at 2 months after completion of neoadjuvant treatment (standard of care since the GRECCAR2 trial).
  Arms: Control: Standard assessment of tumor response (validated in the GRECCAR 2 trial - Lancet 2017)
Other: Follow-up — Every 3 months for 2 years, then every 6 months for the third year

SUMMARY:
The adoption of total mesorectal excision (TME) has standardized rectal cancer surgery and improved oncological outcomes. In locally advanced rectal cancer, neoadjuvant radio chemotherapy (NACRT) has further improved oncological benefit. Although these strategies result in good 5-year disease-free survival rates, they are associated with significant morbidity, in particular permanent long-term bowel, urinary and sexual dysfunction. In rectal cancer management, the main objective of organ preservation is to avoid or reduce morbidity and impact on quality of life after rectal resection, without compromising oncological outcomes.

The aim of this project is to evaluate the efficacy of a defined response monitoring program, including a shared decision process, as a strategy for assessing tumor response in locally advanced rectal cancer after neoadjuvant therapy.

This is a national, phase III, randomized, open-label, multicenter clinical trial comparing the tumor response monitoring program with shared decision-making, versus standard tumor response assessment in organ preservation strategies in rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 to 80
* Histologically proven lieberkuhnian adenocarcinoma with MSS status ;
* Patient who has or is due to receive neoadjuvant treatment (4 to 6 courses of (m)FOLFIRINOX or FOLFOX chemotherapy + CAP 50 radiochemotherapy or CAP 50 radiochemotherapy alone);
* BEFORE any neoadjuvant treatment:

  * Tumor classified T2T3 (on MRI)
  * N0-N1 (≤ 3 positive lymph nodes * or size ≤ 8 mm) (on MRI)
  * * positive node = node size > 5 mm minor axis and/or morphologically suspicious appearance Tumor size ≤4 cm (ON MRI)
  * No distant metastasis (M0)_ TAP scan or PET scan
  * ≤ 8 cm from anal margin (On MRI) (Clinical examination*)

    *if the clinical examination is not possible, then the source data is that of the MRI.
  * No invasion of the anal canal and/or sphincters (internal and external) (On MRI)
* Operable patient
* Ability to comply with the protocol and follow-up appointments (repeated assessment consultations and close follow-up if randomized to the Experimental Group);
* Person affiliated with or benefiting from a social security scheme;
* Free and informed consent signed by the patient.

Exclusion Criteria:

* Patients with a history of chemotherapy or pelvic irradiation (excluding neoadjuvant treatment)
* Contraindication to pelvic MRI
* Patients with MSI status undergoing immunotherapy
* Other concomitant cancer or history of cancer within 5 years, with the exception of carcinoma in situ of the cervix or basal cell or squamous cell skin carcinoma or any other carcinoma in situ, considered cured
* Women who are pregnant, likely to become pregnant, or who are breast-feeding;
* Person under guardianship, curatorship or safeguard of justice, or person deprived of liberty.
* Unable to undergo medical follow-up for geographical, social or psychological reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Organ preservation rate | 2 years after the start of neoadjuvant treatment
  An organ-preserving patient is defined as a patient who has not undergone rectal resection.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France